CLINICAL TRIAL: NCT03557346
Title: Objective Verification of Physiologic Changes During Accommodation Under Binocular, Monocular, and Pinhole Conditions
Status: Completed | Type: Observational
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, Hong Hyun Park, Resident, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Other Study IDs: CAUHOphthalmology
Record Dates: First submitted 2018-05-22; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Accommodation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: the WAM-5500 binocular autorefractor/keratometer (Grand Seiko Co. Ltd., Hiroshima, Japan) — : Subjects underwent a basic ophthalmic examination and the accommodative response to refractive stimuli was measured. Refractive stimuli were given at 0.25 diopters (D) (4 m distance), 2D (50 cm), 3D (33 cm), and 4D (25 cm) and stimulation was applied with the eyes in binocular, monocular (dominant eye, non-dominant eye, ipsilateral, and contralateral), and pinhole conditions. In addition, changes in the astigmatic value and direction of the astigmatism axis under binocular stimulus were evaluated.

SUMMARY:
The investigators believe that this simple, clear, and objective study may be a great help in understanding the accommodative response during various accommodative stimulation conditions.

DETAILED DESCRIPTION:
The purpose in this study was to investigate physiological changes in accommodative power, pupil diameter, astigmatic value, and axis when visual stimuli were applied under binocular, monocular (dominant eye, non-dominant eye, ipsilateral, and contralateral), and pinhole conditions using the WAM-5500 binocular autorefractor/keratometer (Grand Seiko Co. Ltd., Hiroshima, Japan).

ELIGIBILITY:
Inclusion Criteria:

1. age between 20 and 40 years
2. spherical equivalent (SE) within ± 4.0 diopters (D)
3. correctable distant and near visual acuity by glasses to 20/20
4. normal ocular alignment.

Exclusion Criteria:

1. disturbance of accommodation (e.g., Adie's pupil, Parkinson's disease, accommodative esotropia, accommodative spasm, presbyopia)
2. disorders that can affect accommodation (e.g., history of ocular trauma, previous ocular surgery)
3. disorders that might limit testing accuracy (e.g., corneal pathological features, cataract, glaucoma, vitreous opacity, and retinal abnormalities).

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects who visited the department of ophthalmology in Chung-Ang university hospital for ocular examination
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Accommodative power | Subjects performed this examination while being under binocular, monocular, and pinhole conditions with one week apart in random order after baseline study
  Accommodative powers in diopters were measured using WAM-5500 binocular autorefractor/keratometer
Pupil diameter | Subjects performed this examination while being under binocular, monocular, and pinhole conditions with one week apart in random order after baseline study
  Pupil diameters in millimeters were measured using WAM-5500 binocular autorefractor/keratometer
Astigmatic value and axis change | Subjects performed this examination while being under binocular, monocular, and pinhole conditions with one week apart in random order after baseline study
  Astigamtic value in diopters and axis change in degrees were measured using WAM-5500 binocular autorefractor/keratometer The spherical equivalent (sphere + 1/2 cylinder) was used to assess the response to refractive stimuli. The principal meridian of the cylinder for 0.25D refractive stimulus was set to the baseline axis. For 2D, 3D, and 4D refractive stimuli, vertical movement was determined when the baseline meridian moved to the 90' axis, and it was considered horizontal movement when it moved to the 0' or 180' axis.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Park H, Park IK, Shin JH, Chun YS. Objective Verification of Physiologic Changes during Accommodation under Binocular, Monocular, and Pinhole Conditions. J Korean Med Sci. 2019 Jan 21;34(4):e32. doi: 10.3346/jkms.2019.34.e32. eCollection 2019 Jan 28. PMID 30686953